CLINICAL TRIAL: NCT02121067
Title: Intrauterine Contraceptive Insertion at Two-weeks Postpartum: A Study of Acceptability and Short-term Outcomes
Brief Title: LNG-IUS at 2 Weeks Postpartum
Acronym: LNG-IUS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 14-0202
Record Dates: First submitted 2014-03-24; First posted 2014-04-23 (Estimated); Results first posted 2017-06-01 (Actual); Last update posted 2017-08-24 (Actual); Status verified 2017-07

CONDITIONS: Contraception; Malposition of Intrauterine Contraceptive Device
Keywords: postpartum; contraception; intrauterine device; intrauterine system; mirena; uterine involution
MeSH Terms: interventions — Levonorgestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LNG-IUS placed at 2 weeks postpartum (Experimental): Enrolled women will have the LNG-IUS placed at two-weeks (14-20 days) postpartum
  Interventions: Drug: Levonorgestrel Intrauterine System (LNG-IUS)

INTERVENTIONS:
Drug: Levonorgestrel Intrauterine System (LNG-IUS) — The LNG-IUS will be inserted at two-weeks postpartum (day 14-20 postpartum) in all 50 women enrolled
  Other Names: Mirena

SUMMARY:
This is a study of 50 postpartum women interested in having the Mirena® LNG-IUS placed for contraception. The Mirena® is an FDA approved intrauterine contraceptive device that provides contraception for 5 years with excellent effectiveness. Women enrolled in this study will only have the Mirena® placed at two-weeks postpartum (day 14-20 postpartum). The participants will be followed at 6-weeks and 6-months postpartum for study visits to evaluate for satisfaction, symptoms, expulsion, and perforation. The study will be completed at six-months postpartum, and participants will be able to keep their LNG-IUS following study completion.

ELIGIBILITY:
Inclusion Criteria:

1. Desiring a LNG-IUS
2. Postpartum, ages 18-45 who deliver at a gestational age > 32 weeks, delivery can be via cesarean or vaginal delivery
3. Following a viable, singleton pregnancy
4. Willing to return to UNC for their LNG-IUS insertion and study follow-up
5. Who plan to stay in the UNC area for 6 months and willing to return to UNC for 3 visits
6. Fluent in English or Spanish
7. At risk of repeat pregnancy (i.e. excluding those who had tubal sterilization)

Exclusion Criteria:

1. No genital bleeding of unknown etiology
2. No personal history of known or suspected breast carcinoma
3. No 4th degree vaginal laceration at time of delivery
4. No documented uterine rupture during delivery
5. No active liver disease (resolved pre-eclampsia may enroll)
6. No evidence of vaginal, cervical or uterine infection at time of LNG-IUS insertion
7. No history of postpartum endometritis treated with antibiotics or a postpartum readmission for a dilation and curettage
8. No pre-existing contraindication to a LNG-IUS as determined by the CDC's Medical Eligibility Criteria (MEC) category 3 or 4
9. Not currently incarcerated
10. No known congenital or acquired uterine anomaly, including fibroids that distort the uterine cavity
11. No suspected hypersensitivity or contraindication to the LNG-IUS
12. With any other condition or circumstance that the PI determines could cause an adverse event or interfere with completing the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2014-09; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew L Zerden, MD, MPH, Principal Investigator — UNCH; Gretchen S Stuart, MD, Study Director — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Zerden ML, Stuart GS, Charm S, Bryant A, Garrett J, Morse J. Two-week postpartum intrauterine contraception insertion: a study of feasibility, patient acceptability and short-term outcomes. Contraception. 2017 Jan;95(1):65-70. doi: 10.1016/j.contraception.2016.08.005. Epub 2016 Aug 20. PMID 27554014

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LNG-IUS Placed at 2 Weeks Postpartum
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | LNG-IUS Placed at 2 Weeks Postpartum
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 50
  >=65 years | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 30 [24 to 36]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Would Recommend the LNG-IUS to a Friend at 6-months Postpartum.
Description: A dichotomous, yes/no answer to the following question "Would you recommend Mirena placement at two-weeks postpartum to a friend?"
Time Frame: 6 months postpartum
Population: Of the 50 participants who enrolled, only 43 were available at 6 months postpartum to provide data for the first primary outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | LNG-IUS Placed at 2 Weeks Postpartum
Number analyzed (Participants) | 43
Participants | 40

2. Primary Outcome: Number of Participants Who Enrolled and Were Able to Have a Successful LNG-IUS Insertion in the 2 Week (Day 14-20) Postpartum Period.
Description: Was the LNG-IUS successfully placed in the study period, as determined by whether the participant had an LNG-IUS placed on the day of insertion?
Time Frame: Day 14-20 postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | LNG-IUS Placed at 2 Weeks Postpartum
Number analyzed (Participants) | 50
Participants | 50

3. Secondary Outcome: Number of Participants With Expulsion (Complete or Partial) of LNG-IUS at Six-months.
Description: Expulsion will be defined as any of the following (1) patient report that the LNG-IUS came out, (2) ultrasound evaluation that demonstrates the LNG-IUS is not intrauterine (3) ultrasound or clinical evaluation that demonstrates the majority of the LNG-IUS is located in the cervix.
Time Frame: 6 months postpartum
Population: Of the 50 participants who enrolled and had an LNG-IUS placed at 2 weeks postpartum, only 43 were available at 6 months postpartum to provide data for expulsion.
Measure: Count of Participants; unit: Participants
Arm/Group | LNG-IUS Placed at 2 Weeks Postpartum
Number analyzed (Participants) | 43
Participants | 2

ADVERSE EVENTS:
Arm/Group | LNG-IUS Placed at 2 Weeks Postpartum
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes